CLINICAL TRIAL: NCT02178527
Title: A Podiatry Intervention to Reduce Falls in Care Home Residents: Development, Feasibility and Acceptability Study With Exploratory Randomised Controlled Trial
Brief Title: Podiatry Intervention to Reduce Falls in Elderly Care Trial (PIRFECT)
Acronym: PIRFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Stirling (Other); La Trobe University (Other); University of Toronto (Other); University of Dundee (Other)
Responsible Party: Principal Investigator, Gavin Wylie, Principle Investigator, NHS Tayside
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010GR10; CZH/4/701 (Other Grant/Funding Number: Chief Scientist Office, Scottish Goverment)
Record Dates: First submitted 2014-06-17; First posted 2014-06-30 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Accidental Falls
Keywords: Geriatrics; Accidental Falls; Podiatry; Exercise Therapy; Orthotic Devices; Foot
MeSH Terms: interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mulitfaceted podiatry Intervention (Experimental): Foot and ankle exercises, foot orthoses, footwear provision
  Interventions: Other: Foot and ankle exercises, foot orthoses, footwear provision
- Usual podiatry care (Placebo Comparator): Continued provision of usual NHS (National Health Service) podiatry care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Foot and ankle exercises, foot orthoses, footwear provision — Participants in the intervention group will receive orthoses and footwear as part of the study. The research team will train care home staff in the provision of foot and ankle exercises. The exercise protocol states that exercises will be carried out 3 times per week for 12 weeks.
  Arms: Mulitfaceted podiatry Intervention
Other: Usual Care — Usual general podiatry care provded by UK National Health Service
  Arms: Usual podiatry care

SUMMARY:
This is an exploratory pilot Randomised Controlled Trial (RCT) to investigate the effects of a multifaceted podiatry intervention designed to reduce falls in care homes. The investigators hypothesise that the intervention will reduce the high falls rates present in care homes for older people, compared to usual care.

The results will inform the sample size calculation for a full-scale definitive RCT

DETAILED DESCRIPTION:
Background: Falls are a problem in care homes where it is estimated that half of all residents will fall at least once in a year. There is now strong empirical evidence that weakness of the foot muscles and painful foot problems such as corns and/or callus are a contributing factor to falls in this population. These problems are common and reversible; however there have been no trials of podiatry interventions that address these problems to establish whether or not this approach can be effective at reducing falls in care home populations.

Methods: Care home residents meeting the inclusion criteria will be assigned to receive either the intervention (specific foot and ankle exercises, orthoses, footwear). We will then conduct an exploratory randomised controlled trial (RCT) with the aim of acquiring data that will inform the design of a subsequent full scale RCT. The groups will then be compared on a number of balance and falls related outcomes.

Main Outcome: The results will indicate the effect size to allow a sample size calculation for a later definitive trial to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 65 Years or older permanently living in care homes for older people
* One or more falls in the previous year.
* Foot problem that is within the scope of podiatry care

Exclusion Criteria:

* Residents who are terminally unwell or too frail to be included
* Residents who are only able to mobilise with the use of a wheelchair
* Temporary residents (for example, those in respite care)
* Unable to provide informed consent
* Lower limb Amputees

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in falls rate | 3 months from baseline measures, 6 months from baseline, 9 months from baseline
  A fall will be defined as "an unexpected event in which the participant comes to rest on the ground, floor, or lower level"

SECONDARY OUTCOMES:
Functional Balance: Berg Balance Scale | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline
Mobility: Timed up and go test | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline
Physical Functioning: Barthel Index | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline
Health Related Quality of Life: EQ-5D | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline
Foot and Ankle Strength | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline
  Measured via hand held dynamometry
Falls efficacy: Nursing home falls self efficacy scale | Baseline, 3 months from baseline measures, 6 months from baseline, 9 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gavin H Wylie, MSc, Principal Investigator — NHS (National Health Service) Tayside / University of Dundee
Locations (9):
- United Kingdom (9):
  - Glencairn House Care Home, Auchterarder
  - Ancaster Care Home, Crieff
  - Harestane Care Home, Dundee
  - Janet Brougham House, Dundee
  - Balcarres Care Home, Dundee
  - Orchar Care Home, Dundee
  - Rivendell Care Home, Dunkeld
  - Craigieknowes Care Home, Perth
  - Kincarrathie House Care Home, Perth

REFERENCES:
- [Derived] Wylie G, Menz HB, McFarlane S, Ogston S, Sullivan F, Williams B, Young Z, Morris J. Podiatry intervention versus usual care to prevent falls in care homes: pilot randomised controlled trial (the PIRFECT study). BMC Geriatr. 2017 Jul 12;17(1):143. doi: 10.1186/s12877-017-0541-1. PMID 28701161